CLINICAL TRIAL: NCT06998108
Title: A Multicenter, Randomized, Controlled, Double-blind Phase III Clinical Study of BEBT-209 in Combination With Fulvestrant Versus Placebo in Combination With Fulvestrant for the Treatment of HR+/HER2- Locally Advanced or Metastatic Breast Cancer in Patients With Disease Progression After Prior Endocrine Therapy
Brief Title: Study of BEBT-209 in Combination With Fulvestrant Versus Placebo in Combination With Fulvestrant in Patients With HR+/HER2- Locally Advanced or Metastatic Breast Cancer Who Have Progressed After Prior Endocrine Therapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BeBetter Med Inc (Industry)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GBMT-209-P04
Record Dates: First submitted 2025-05-29; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: HR+/HER2- Locally Advanced, Metastatic Breast Cancer
Keywords: BEBT-209; Efficacy; Safety
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BEBT-209+ Fulvestrant (Active Comparator): BEBT-209 75 mg twice daily on days 1-21 in combination with fulvestrant 500 mg once daily (day 1 and day 15 of cycle 1; subsequent cycles: day 1).
  Interventions: Drug: BEBT-209 capsules; Drug: Fulvestrant Injection
- BEBT-209 Placebo + Fulvestrant (Placebo Comparator): Placebo 75 mg twice daily on days 1-21 in combination with fulvestrant 500 mg once daily (day 1 and day 15 of cycle 1; subsequent cycles: day 1).
  Interventions: Drug: BEBT-209 Placebo capluses; Drug: Fulvestrant Injection

INTERVENTIONS:
Drug: BEBT-209 capsules — Oral, 75 mg per dose, twice daily, in a 28-day cycle. Continuous dosing from day 1 to day 21, followed by a rest period from day 22 to day 28.
  Other Names: BEBT-209
  Arms: BEBT-209+ Fulvestrant
Drug: BEBT-209 Placebo capluses — Oral, 75 mg per dose, twice daily, in a 28-day cycle. Continuous dosing from day 1 to day 21, followed by a rest period from day 22 to day 28.
  Arms: BEBT-209 Placebo + Fulvestrant
Drug: Fulvestrant Injection — 500 mg intramuscular injection, with a 28-day treatment cycle. Administration on day 1 and day 15 of the first cycle, and then on day 1 of each subsequent cycle.

SUMMARY:
This study is a randomized, double-blind, multicenter, placebo-controlled Phase III clinical trial designed to evaluate the efficacy and safety of BEBT-209 in combination with fulvestrant in patients with HR+/HER2- locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
This study plans to enroll 330 eligible female patients with locally advanced or metastatic breast cancer. All eligible patients will be randomly assigned to the treatment group or the control group in a 2:1 ratio. The following two factors will be used for stratification: 1) visceral metastasis (yes or no); 2) menopausal status (postmenopausal; premenopausal or perimenopausal). The study consists of a screening period, a treatment period, and a follow-up period. It aims to evaluate the efficacy and safety of BEBT-209 in combination with fulvestrant versus placebo in combination with fulvestrant in patients with HR+/HER2- locally advanced or metastatic breast cancer who have experienced disease progression after prior endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 years or older who are postmenopausal or premenopausal/perimenopausal, and meet one of the following criteria: previous bilateral oophorectomy, or age ≥60 years; or age <60 years with natural menopause (defined as spontaneous cessation of regular menstruation for at least 12 consecutive months without other pathological or physiological causes), and estradiol (E2) and follicle-stimulating hormone (FSH) levels in the postmenopausal range; or premenopausal or perimenopausal women willing to receive luteinizing hormone-releasing hormone (LHRH) agonist therapy during the study period.
2. Patients with histologically confirmed HR+/HER2- breast cancer (based on the most recent test results from either recurrent/metastatic lesion tissue samples or prior primary lesion tissue samples): a) ER+ and/or PR+ is defined as ≥10% of tumor cells showing positive staining for ER/PR; b) HER2- is defined as an immunohistochemistry(IHC) score of 0 or 1+, or a fluorescence in situ hybridization(FISH) ratio of HER2/CEP17 less than 2.0, or HER2 gene copy number less than 4.
3. Evidence of focal recurrence or metastasis, not suitable for curative surgery or radiotherapy, and without clinical indications necessitating chemotherapy.
4. Previous endocrine therapy must meet one of the following criteria: a) progression during or within 12 months after discontinuation of adjuvant endocrine therapy (with an aromatase inhibitor [aromatase inhibitor or selective estrogen receptor modulator such as tamoxifen, toremifene, etc.); b) progression during or within 1 month after discontinuation of endocrine therapy for first recurrence or metastasis.
5. Patients are allowed to have received no more than one line of chemotherapy during the recurrence or metastatic phase.
6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
7. Presence of measurable lesions according to response evaluation criteria in solid tumors (RECIST) 1.1 criteria or bone metastases only (including lytic or mixed lesions).
8. Adequate organ and marrow function, defined as follows: absolute neutrophil count (ANC) ≥1.5×10⁹/L (without use of growth factors within 14 days); platelets ≥100×10⁹/L (without corrective treatment within 7 days); hemoglobin ≥90 g/L (without corrective treatment within 7 days); serum creatinine ≤1.5 times the upper limit of normal (ULN) or estimated creatinine clearance ≥60 mL/min; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 times the ULN (≤5 times the ULN for patients with liver metastases); total serum bilirubin (TBIL) ≤2.5 times the ULN; 12-lead electrocardiogram: Fridericia-corrected QT interval (QTcF) < 470 msec (for females).
9. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose of study drug and must be willing to use a medically accepted and highly effective method of contraception from the time of signing the informed consent form, throughout the study period, and for 1 year after the last administration of the study drug.
10. All acute toxicities from prior anti-tumor therapy must have resolved to grade 0-1 (according to national cancer institute(NCI) common terminology criteria for adverse events(CTCAE) version 5.0) or to the levels specified in the inclusion/exclusion criteria. Exceptions include alopecia and other toxicities deemed by the investigator to pose no safety risk to the patient.
11. The patient has provided written informed consent and is willing and able to comply with the planned visits, study treatment schedule, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Patients who are deemed by the investigator to be unsuitable for endocrine therapy, including those with symptomatic, visceral metastatic disease, or those at risk of life-threatening complications in the short term (including patients with uncontrollable effusions [pleural, pericardial, peritoneal] despite drainage or other measures, pulmonary lymphangitis, or more than 50% liver involvement).
2. Known uncontrolled or symptomatic active central nervous system (CNS) metastases, characterized by clinical symptoms, brain edema, spinal cord compression, carcinomatous meningitis, leptomeningeal disease, and/or progressive growth; patients with a history of CNS metastases or spinal cord compression may be eligible if they have received definitive treatment and have been clinically stable for 4 weeks after discontinuation of anticonvulsants and corticosteroids prior to the first dose of study drug.
3. Previous treatment with fulvestrant, everolimus, or CDK4/6 inhibitors.
4. From the end of the last treatment to the first dose: underwent surgical or radiation therapy within 14 days prior to the first dose and has not fully recovered from the treatment; received chemotherapy, any investigational drug, or other anti-cancer therapy within 14 days or within five half-lives of the therapeutic agent prior to the first dose (whichever is longer is acceptable for enrollment).
5. A diagnosis of any other malignancy within 3 years prior to randomization, with the exception of non-melanoma skin cancer (basal cell or squamous cell carcinoma) or cervical carcinoma in situ that has been treated with curative intent.
6. Infection with human immunodeficiency virus (HIV) or known acquired immune deficiency syndrome (AIDS); active hepatitis B (patients positive for hepatitis B surface antigen [HBsAg] and with hepatitis B virus DNA [HBV-DNA] levels above the ULN of the local laboratory). Patients with HBV DNA levels above the ULN of the local laboratory are permitted to receive antiviral therapy prior to screening, and may be enrolled once viral copies are reduced below the ULN, but must continue antiviral therapy for hepatitis B during the study; hepatitis C (positive for hepatitis C virus antibody and with HCV RNA levels above the ULN of the local laboratory); or co-infection with both hepatitis B and hepatitis C.
7. Within 6 months prior to randomization, the following conditions have occurred: myocardial infarction, severe/unstable angina, heart failure of NYHA Class II or higher, persistent arrhythmia of Grade ≥2 (according to NCI CTCAE Version 5.0), atrial fibrillation of any grade, coronary/peripheral artery bypass grafting, symptomatic congestive heart failure, cerebrovascular accident (including transient ischemic attack), or symptomatic pulmonary embolism.
8. Severe infection within 4 weeks prior to the first dose (e.g., requiring intravenous antibiotics, antifungal, or antiviral therapy according to clinical practice guidelines), or unexplained fever >38.5℃ during the screening period or prior to the first dose.
9. Inability to swallow, intestinal obstruction, or other factors that may affect the intake and absorption of medication.
10. Known coagulation abnormalities; or use of anticoagulant therapy prior to intramuscular injection of fulvestrant or LHRH agonist (goserelin).
11. Known allergy to fulvestrant, LHRH agonist (goserelin), BEBT-209/placebo, or any of their excipients.
12. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
13. Known history of abuse of psychoactive substances or drug addiction.
14. Poorly controlled diabetes mellitus as judged by the investigator.
15. Uncontrolled hypertension as judged by the investigator.
16. Presence of other severe physical or psychiatric conditions or laboratory abnormalities that may increase the risk of participation in the study, interfere with the study results, or render the patient unsuitable for participation in the study as judged by the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
PFS assessed by the Independent Imaging Review Committee | Up to 56 weeks
  Progression free survival (PFS) assessed by the Independent Imaging Review Committee

SECONDARY OUTCOMES:
PFS assessed by investigators | Up to 56 weeks
  Progression free survival assessed by investigators
OS | Up to 56 weeks
  Overall Survival
ORR | Up to 56 weeks
  Overall Objective Response
CBR | Up to 56 weeks
  Clinical Benefit Rate
DOR | Up to 56 weeks
  Duration of Response
Occurrence of Adverse Events (AEs) | Up to 36 months
  Occurrence of AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE V5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, Ph.D, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China